CLINICAL TRIAL: NCT04522661
Title: Early Vitrectomy and Intravitreal Antibiotics for Post-operative Exogenous Endophthalmitis: A Feasibility Multicentre Randomised Controlled Trial (EVIAN Study)
Brief Title: A Feasibility Randomised Controlled Trial of Early Vitrectomy for Post-operative Exogenous Endophthalmitis
Acronym: EVIAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: University College, London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUQM1006
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Endophthalmitis Postoperative Acute
Keywords: vitrectomy; intravitreal antibiotics
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Vitrectomy Group (Experimental): Vitrectomy surgery plus intravitreal antibiotics
  Interventions: Procedure: Vitrectomy; Procedure: Intravitreal antibiotics
- Control Group (Active Comparator): Intravitreal antibiotics
  Interventions: Procedure: Intravitreal antibiotics

INTERVENTIONS:
Procedure: Vitrectomy — Vitrectomy within 48 hours of randomisation
  Arms: Early Vitrectomy Group
Procedure: Intravitreal antibiotics — Intravitreal Antibiotics at 48 hours

SUMMARY:
This randomised clinical trial will explore the feasibility and acceptability of carrying out early vitrectomy surgical treatment compared to standard treatment in acute endophthalmitis. We will investigate the effectiveness of early vitrectomy plus intravitreal antibiotics compared to standard care intravitreal antibiotic injections in the management of postoperative exogenous endophthalmitis. This is a feasibility trial that will evaluate the expected effect size with which to inform the design of a definitive randomized trial of this question.

DETAILED DESCRIPTION:
The EVIAN Study is a multicentre, feasibility, randomised controlled trial to evaluate the effect of early vitrectomy surgery on acute endophthalmitis.

Patients with postoperative exogenous endophthalmitis following any ocular surgery/procedure/injection intervention will be recruited at 48 hours following initial presentation.

Patients with vision of 35 ETDRS letters or better are ineligible for the trial, and would continue on standard of care management. Patients with vision of worse than 35 ETDRS letters will be eligible for the study. At the 48-hour time-point, eligible patients will be randomised in a 1:1 ratio.

The treatment group will undergo vitrectomy within 48 hours of randomisation. The control group will have continued intravitreal antibiotic eye injections according to local protocols. If the vision reaches perception of light, then a vitrectomy surgery would be considered as part of standard of care at 12-15 days. Follow up will be for 6 months in both groups.

Visual acuity, funds photography, B-scan ultrasound, and optical coherence tomography (OCT) scanning will be performed from baseline until the final follow-up at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patient over 18 years of age
* Patient has capacity to give informed consent
* Patient has not previously been enrolled in this study in regards to their other eye
* Diagnosis of postoperative endophthalmitis at any time-point following an ocular surgery/procedure/injection
* Patient is healthy to undergo vitrectomy surgery
* Symptomatic Visual loss attributable to POE
* Best corrected visual acuity worse than 35 ETDRS letters, including CF, HM and POL vision

Exclusion Criteria:

* Patient suffered a major thromboembolic event within the past 3 months as (defined as TIA, Stroke, or MI)
* Known adverse reaction to intravitreal antibiotics (amikacin/vancomyin/cephalosporins)
* Blood pressure greater than 200 systolic or 100 diastolic
* Any other condition that in the opinion of the investigator would preclude participation in the study (such as unstable medical status or severe disease that would make it difficult for the patient to be able to complete the study)
* The patient will use an investigational drug during the study
* History of optic atrophy in the study eye
* Corneal oedema/haze that would prevent visualisation of fundus to perform vitrectomy surgery
* Patient over the age of 95 who present with POE should immediately be placed on the pre-screening log as ineligible

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Patient recruitment | Trial study period (Week 1 to Week 104)
  Number of participants

SECONDARY OUTCOMES:
Distance Best Corrected Visual Acuity change from baseline | Trial study period (Week 1 to Week 24)
  Early Treatment Diabetic Retinopathy Study (ETDRS) letters

CONTACTS AND LOCATIONS:
Overall Officials: Mahi MK Muqit, PhD FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results to be reported in an International Committee of Medical Journal Editors journal after deidentification (text, tables, figures, and appendices)
Supporting Information: SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. The access should only be for individual participant data meta-analysis.

REFERENCES:
- [Background] Results of the Endophthalmitis Vitrectomy Study. A randomized trial of immediate vitrectomy and of intravenous antibiotics for the treatment of postoperative bacterial endophthalmitis. Endophthalmitis Vitrectomy Study Group. Arch Ophthalmol. 1995 Dec;113(12):1479-96. PMID 7487614
- [Background] Negretti GS, Chan W, Pavesio C, Muqit MMK. Vitrectomy for endophthalmitis: 5-year study of outcomes and complications. BMJ Open Ophthalmol. 2020 Mar 24;5(1):e000423. doi: 10.1136/bmjophth-2019-000423. eCollection 2020. PMID 32258421
- [Background] Busbee BG, Recchia FM, Kaiser R, Nagra P, Rosenblatt B, Pearlman RB. Bleb-associated endophthalmitis: clinical characteristics and visual outcomes. Ophthalmology. 2004 Aug;111(8):1495-503; discussion 1503. doi: 10.1016/j.ophtha.2004.01.028. PMID 15288977
- [Derived] Muqit MMK, Pavesio C, Boston H, Sriharan K, Wang Y, Pizzo E, Cobb S, Spink C, Bainbridge J. A Randomised Controlled Trial of Early Vitrectomy and Intravitreal Antibiotics for Post-operative Exogenous Endophthalmitis (EVIAN study): study protocol for a feasibility trial. NIHR Open Res. 2023 Sep 28;3:47. doi: 10.3310/nihropenres.13469.1. eCollection 2023. PMID 39139269